CLINICAL TRIAL: NCT05777642
Title: in Vivo Double-blind, Randomized, Placebo Controlled, Crossover Investigation of the Effect of Oral Administration of an Oxygen-nanobubble Drink on the Exercise Performance in Elite Athletes
Brief Title: Oxygen Nanobubble Drink Impact on Exercise in Elite Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: R83003/RE001
Record Dates: First submitted 2023-02-13; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen Nanobubble First (Experimental): In this arm, the oxygen nanobubbles drink will be provided as the first drink. The oxygen nanobubbles mixture will be mixed with water and oxygenated and provided as a one-time 200ml drink 10 minutes before the start of the 2000m row.
  The placebo will be provided as the second drink, 2-4 days after the first drink. The placebo mixture will be mixed with water and oxygenated and provided as a one-time 200ml drink 10 minutes before the start of the 2000m row.
  Interventions: Dietary Supplement: Oxygen Nanobubble; Dietary Supplement: Placebo
- Placebo First (Placebo Comparator): In this arm, the placebo drink will be provided as the first drink. The placebo mixture will be mixed with water and oxygenated and provided as a one-time 200ml drink 10 minutes before the start of the 2000m row.
  The oxygen nanobubbles will be provided as the second drink, 2-4 days after the first drink. The oxygen nanobubbles mixture will be mixed with water and oxygenated and provided as a one-time 200ml drink 10 minutes before the start of the 2000m row.
  Interventions: Dietary Supplement: Oxygen Nanobubble; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oxygen Nanobubble — This contains oxygenated nanobubbles made from lecithin and natural flavourings (Liquorice, glycerol, and citric acid)
Dietary Supplement: Placebo — This does not contain nanobubbles and is made from natural flavourings (Liquorice, glycerol, and citric acid)

SUMMARY:
Although the primary organ of gas exchange is the lung, it has been recognized for some time that other organs have a potential role in gas exchange. There is emerging evidence that the gastrointestinal tract may have the capacity to act as an organ of gas exchange.

Several recent studies in both animals and humans have indicated that orally administered oxygenated nanobubbles is a safe intervention that can improve tissue oxygenation. Oxygen nanobubbles can reduce the hypoxia in tumours when injected, in conjunction with sonodynamic therapy. In mice, researchers have shown a reduction in tumour hypoxia and improved response to sonodynamic therapy occurs even when the oxygen nanobubbles are orally administered.

This will be an in vivo randomized, double-blinded, cross-over, placebo-controlled study consisting of rowers. By measuring the time taken by participants to complete a 2000m row after consuming an Oxygen nanobubbles drink, and a placebo drink, the investigators will evaluate the efficacy of the nanobubbles on the exercising ability of the participant.

DETAILED DESCRIPTION:
Although the primary organ of gas exchange is the lung, it has been recognized for some time that other organs have a potential role in gas exchange. There is emerging evidence that the gastrointestinal tract may have the capacity to act as an organ of gas exchange. Several animal studies have demonstrated that oxygen (delivered as a gas and within enriched water) is capable of diffusing through the mucosa of the colon, peritoneum and stomach resulting in elevated oxygen tension in the splanchnic circulation (hepatic portal vein, arterial and venous mixed blood) and increased blood flow (portal venous blood flow). One MRI study has demonstrated that orally administered oxygen-supersaturated water causes a significant increase in the luminal oxygen concentration in both the oral cavity and the stomach, despite a low amount of oxygen added to the overall oxygen balance of the body.

Several recent studies in both animals and humans have indicated that orally administered oxygenated nanobubbles is a safe intervention that can improve tissue oxygenation. Oxygen nanobubbles can reduce the hypoxia in tumours when injected, in conjunction with sonodynamic therapy. In mice, researchers have shown a reduction in tumour hypoxia and improved response to sonodynamic therapy occurs even when the oxygen nanobubbles are orally administered. A study of male cyclists also showed that ingested oxygen nanobubbles led to an increased power output.

This will be an in vivo randomized, double-blinded, cross-over, placebo-controlled study consisting of rowers. By measuring the time taken by participants to complete a 2000m row after consuming an Oxygen nanobubbles drink, and a placebo drink, the efficacy of the nanobubbles on the exercising ability of the participant will be evaluated. This will be supplemented with a comparison of a pre-intervention and post-intervention validated Rate of Perceived Exertion (RPE) breathlessness questionnaire and measurement of blood lactate and glucose, blood gases, respiratory gas exchange and heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the research
* Participant is 18+ years of age
* Not currently taking any medications (except the contraceptive pill)
* The participant must be a competitive rower, with an estimated 2000m time of ≤6:30 minutes for males, and ≤ 8 minutes for females.
* The participant agrees to abstain from tobacco and nicotine products 24 hours before each visit.
* The participant agrees to abstain from alcohol 24 hours before each visit.
* The participant is, in the opinion of the investigator, healthy on the basis of a self-reported medical history, vital signs.
* The participant has no active disease process that could interfere with endpoints.
* Available for the duration of the study.
* The participant is not taking regular medications (including NSAIDs such as ibuprofen) that could interfere with endpoints measured and/or influence gastrointestinal permeability and led to gastrointestinal symptoms.
* The participant has not taken dietary/nutritional supplements in the preceding 2 weeks.
* The participant is not following a weight reducing diet.
* The participant is willing not to undertake strenuous or unaccustomed physical exercise for at least 24 hours prior to screening and study visits.

Exclusion Criteria:

* Participants with a history of smoking in the previous 30 days
* Participants that are allergic or intolerant towards: Liquorice, Lecithin derived from soya or sunflower, Citric acid, Glycerol
* Clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or haematological disease or abnormality, as determined by the self-reported health questionnaire.
* History of alcohol, narcotic, benzodiazepine, or other substance abuse or dependence within the 12 months preceding study visit 1.
* Currently participating in another study with an investigational or non-investigational drug or device, or has participated in another clinical study within the 2 months preceding study visit 1 (based on participant's self report).
* Any condition that, in the investigator's opinion, compromises the participant's ability to meet protocol requirements or to complete the study.
* Participant is pregnant and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2024-05-18 (Estimated); Study Completion 2024-06-18 (Estimated)

PRIMARY OUTCOMES:
2000m Row Time | 7 days
  Time taken to complete 2000m Row

SECONDARY OUTCOMES:
Heart Rate | 7 days
  Changes in the Heartrate before and after the 2000m Row with the oxygen nanobubbles drink compared with the placebo drink
Peripheral Oxygen Saturation (SpO2) | 7 days
  Changes in the Oxygen Saturation (SpO2) before and after the 2000m Row with the oxygen nanobubbles drink compared with the placebo drink.
  The oxygen saturation (SpO2) will be measured by a pulse oximeter on a scale of 0-100%.
Rate of Perceived Exertion | 7 days
  Changes in the Rate of Perceived Exertion before and after the 2000m Row with the oxygen nanobubbles drink compared with the placebo drink.
  This uses the Borg scale from 6-20, where 6 indicates light exertion, and 20 indicates maximal exertion
Blood Lactate | 7 days
  Changes in the blood lactate before and after the 2000m Row with the oxygen nanobubbles drink compared with the placebo drink.
Blood Glucose | 7 days
  Changes in the blood glucose before and after the 2000m Row with the oxygen nanobubbles drink compared with the placebo drink.

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Handa, Principal Investigator — University of Oxford

IPD SHARING:
Plan to Share IPD: No